CLINICAL TRIAL: NCT02594904
Title: A Multicenter Study to Evaluate the Efficacy of Yinzhihuang Oral Liquid on Indirect Bilirubin of Neonates With Glucose-6-phosphate Dehydrogenase Deficiency
Brief Title: Efficacy of Yinzhihuang Oral Liquid on Indirect Bilirubin of Neonates With Glucose-6-phosphate Dehydrogenase Deficiency
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Weimin Huang, Chief physician, Southern Medical University, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: whuang201500601
Record Dates: First submitted 2015-10-28; First posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Neonatal Hyperbilirubinemia
Keywords: G6PD Deficiency; Neonatal Hyperbilirubinemia; Yinzhihuang Oral Liquid; Indirect Bilirubin
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Glucosephosphate Dehydrogenase Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- G-6-PD normal group (Experimental): Drug: Yinzhihuang Oral Liquid, dose: 3ml each time, 3 times every day, during the period, measuring bilirubin from skin one time every 24 hours.
  Interventions: Drug: Yinzhihuang Oral Liquid
- G-6-PD mild deficiency group (Experimental): Drug: Yinzhihuang Oral Liquid, dose: 3ml each time, 3 times every day, during the period, measuring bilirubin from skin one time every 24 hours.
  Interventions: Drug: Yinzhihuang Oral Liquid
- G-6-PD moderate deficiency group (Experimental): Drug: Yinzhihuang Oral Liquid, dose: 3ml each time, 3 times every day, during the period, measuring bilirubin from skin one time every 24 hours.
  Interventions: Drug: Yinzhihuang Oral Liquid
- G-6-PD sever deficiency group (Experimental): Drug: Yinzhihuang Oral Liquid, dose: 3ml each time, 3 times every day, during the period, measuring bilirubin from skin one time every 24 hours.
  Interventions: Drug: Yinzhihuang Oral Liquid

INTERVENTIONS:
Drug: Yinzhihuang Oral Liquid — All the four groups will be given same treatment as being described in arm description.
  Other Names: Huarun Yinzhihuang Oral solution

SUMMARY:
Neonatal Glucose-6-phosphate Dehydrogenase(G6PD) Deficiency is one of the significant reason for neonatal hyperbilirubinemia and even irreversible bilirubin encephalopathy.The neonates may be attacked due to acute infection, eating beans or exposure to oxidative drugs, etc.

The main clinical manifestations are hemolytic anemia, and the resulting hyperbilirubinemia. When bilirubin is pretty high in body, bilirubin may spread into brain, and thus cause nervous system damage, and severely affect the prognosis of neonates. Therefore, monitoring and early intervention of jaundice has important significance to prevent further aggravation of jaundice and certain sequelae. Phototherapy and exchange transfusion are mainly suitable methods for severe hyperbilirubinemia, however, patients need to be hospitalized. Yinzhihuang Oral Liquid is a kind of traditional Chinese medicine for jaundice. Many large sample and multicenter clinical studies show that the positive efficacy of Yinzhihuang Oral Liquid in the treatment of neonatal hyperbilirubinemia is exactly confirmed.

The purpose of this study is try to detect the treatment effect of Yinzhihuang Oral Liquid on indirect bilirubin in neonates with G-6-PD enzyme deficiency and neonatal hyperbilirubinemia. Try to provide scientific theories for Yinzhihuang Oral Liquid to treat neonates with G-6-PD enzyme deficiency and neonatal hyperbilirubinemia.

DETAILED DESCRIPTION:
The primary objective is to detect the treatment effect of Yinzhihuang Oral Liquid on indirect bilirubin in neonates with G-6-PD enzyme deficiency and neonatal hyperbilirubinemia. Try to provide scientific theories for Yinzhihuang Oral Liquid to treat neonates with G-6-PD enzyme deficiency and neonatal hyperbilirubinemia.

Study subjects includes neonates with hyperbilirubinemia from five hospitals, who are willing to take Yinzhihuang oral liquid.

Five hospitals are South Hospital of Southern Medical University (primary institute), The Third Affiliated Hospital of Guangzhou medical university, Shenzhen maternal and child health hospital, First Affiliated Hospital of Guangxi Medical University, The maternal and child health hospital of Guangxi Zhuang Autonomous Region Inclusion criteria：

1. Full-term newborns with jaundice after 3-7 days of birth, total bilirubin in serum or transcutaneous bilirubin is between 100umol/L and 257umol/L, and start taking Yinzhihuang oral liquid, dose: 3ml per each time, 3 times per each day, during the period, measuring bilirubin from skin one time every 24 hours;
2. Gestational age≥37 weeks, birth weight≥2.5Kg, Apgar scores≥8;
3. lineal consanguinity are all the native residents from Guangdong or Guangxi;
4. The enzyme activity of G-6-PD will be detected and collected from all the neonates subjects;
5. Informed consents of all the neonates subjects are needed. Exclusion Criteria： (1) Neonates with inherited metabolic diseases; (2) Neonates with congenital malformation of liver and gallbladder; (3) Neonates with asphyxia, hypoxia, acidosis, sepsis, high fever, low temperature, low protein, low blood sugar, etc. which may lead to bilirubin encephalopathy; (4)History of oxidation drug exposure(e.g. honeysuckle bath) Study procedures： Outpatient and inpatient neonates (mainly for cesarean section newborns), with jaundice after 3-7 days of birth, total bilirubin in serum or measuring bilirubin from skin is between 100umol/L and 257umol/L, will be selected. On the first day of jaundice, the G-6-PD enzyme activity will be detected by checking arterial blood, and then start taking Yinzhihuang oral liquid, dose: 3ml each time, 3 times every day, during the period, measuring bilirubin from skin one time every 24 hours.

When the transcutaneous bilirubin is below 100umol/L, stop taking the medication. When bilirubin increases to match the phototherapy indications, the neonates will be transferred to the neonatal department, and continue the Yinzhihuang oral liquid treatment until bilirubin decreasing to normal level.

after the transfer to the ICU still needs to continue to use until the jaundice decreased to normal level.

The neonates 's families have to sign the informed consents before entering the study.

G-6-PD <10.37U /g.H b was diagnosed as a lack of G-6-PD activity. Subgroup: according to the severity of the lack of the activity of the enzyme, it will be divided into 3 groups: mild deficiency: 6.93-10.37U/g.H b; moderate deficiency: 3.47-6.92U/g. Hb; severe deficiency: 0-3.46U/g.H b.

Note: the above criteria can be modified according to the test methods of those five hospitals, and will be uniformed by same final standards.

The normal value of G-6-PD enzyme activity is 2.5-5.8KU/L in our hospital, <2.5KU/L can be diagnosed as lack of G-6-PD enzyme activity. However, there is no certain standards for the definition of mild deficiency, moderate deficiency and severe deficiency in our hospital. It was reported that activity is less than 10% of normal is severe deficiency, less than 10%-60% of normal is moderate deficiency, less than 60% of normal is mild deficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Full-term newborns with jaundice after 3-7 days of birth, total bilirubin in serum or transcutaneous bilirubin is between 100umol/L and 257umol/L, and start taking Yinzhihuang oral liquid, dose: 3ml per each time, 3 times per each day, during the period, measuring bilirubin from skin one time every 24 hours;
2. Gestational age≥37 weeks, birth weight≥2.5Kg, Apgar scores≥8;
3. lineal consanguinity are all the native residents from Guangdong or Guangxi;
4. The enzyme activity of G-6-PD will be detected and collected from all the neonates subjects;
5. Informed consents of all the neonates subjects are needed.

Note: Icterus testers are Minolta 105 type. Measurements of bilirubin are from three location, inluding forehead, chest and abdomen. The value of bilirubin will use the average value from the three location, and the unit is umol / L.

Exclusion Criteria:

1. Neonates with inherited metabolic diseases;
2. Neonates with congenital malformation of liver and gallbladder;
3. Neonates with asphyxia, hypoxia, acidosis, sepsis, high fever, low temperature, low protein, low blood sugar, etc. which may lead to bilirubin encephalopathy;
4. History of oxidation drug exposure(e.g. honeysuckle bath)

Ages: 3 Days to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-04 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
The change(umol/L) from baseline of total bilirubin(umol/L) will be calculated and finalized | Every 24 hours during dosing, for around three days.(Typicall the dosing will be stopped once the bilirubin is below 100umol/L)
  Value of the total bilirubin in serum(umol/L) will be collected and calculated.

SECONDARY OUTCOMES:
The percent change(%) from baseline of total bilirubin(umol/L) will be calculated and finalized | Every 24 hours during dosing, for around three days.(Typicall the dosing will be stopped once the bilirubin is below 100umol/L)
  Value of the total bilirubin in serum(umol/L) will be collected and calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Weimin Huang, Ph.D, Principal Investigator — The South Hospital of Southern Medical University
Locations (1):
- The South Hospital of Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Kaplan M, Hammerman C. Glucose-6-phosphate dehydrogenase deficiency and severe neonatal hyperbilirubinemia: a complexity of interactions between genes and environment. Semin Fetal Neonatal Med. 2010 Jun;15(3):148-56. doi: 10.1016/j.siny.2009.10.007. Epub 2009 Nov 26. PMID 19942489
- [Background] Nkhoma ET, Poole C, Vannappagari V, Hall SA, Beutler E. The global prevalence of glucose-6-phosphate dehydrogenase deficiency: a systematic review and meta-analysis. Blood Cells Mol Dis. 2009 May-Jun;42(3):267-78. doi: 10.1016/j.bcmd.2008.12.005. Epub 2009 Feb 23. PMID 19233695
- [Background] Clinical Research Collaborative Group of Yinzhihuang Oral Solution. [A multicenter randomized controlled study on the efficacy and safety of Yinzhihuang oral solution for the treatment of neonatal indirect hyperbilirubinemia in term newborn infants]. Zhonghua Er Ke Za Zhi. 2011 Sep;49(9):663-8. Chinese. PMID 22176900